CLINICAL TRIAL: NCT00435630
Title: Documenting a Learning Curve and Test-retest Reliability of a Virtual Reality Training Simulator in Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Dennis Fowler, Gerald and Janet Carrus Professor of Clinical Surgical Science (In Surgery), Columbia University
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: AAAA7372
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Education
Keywords: Education; Virtual Reality; Laparoscopic Surgery; Learning Curve

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Completing simulator training sessions
  Interventions: Other: LapSim training

INTERVENTIONS:
Other: LapSim training — complete curriculum training on LapSim surgical simulator

SUMMARY:
The purpose of this study is to determine the learning curve for each of seven tasks in a virtual reality laparoscopic simulator by medical students.

DETAILED DESCRIPTION:
Developing objective methodology for assessing technical skill is paramount to superior surgical training. Alternatives to the traditional apprenticeship model of surgical training are necessary in today's emphasis on cost containment and professional competency.

Metrics are widely employed in virtual environments and provide a yardstick for performance measurement. The current method of defining metrics for medical simulation remains more an art than a science. Many studies have demonstrated that trainees who practice laparoscopic skills in a simulated environment will improve their mastery of those skills when tested in that same environment. Fewer studies have been able to document the learning curve for mastery of tasks in a virtual reality simulator. This study will investigate the learning curve for tasks in a virtual reality laparoscopic simulator.

ELIGIBILITY:
Inclusion Criteria:

* Medical students, years 1 through 4 are eligible.
* No prior clinical experience with laparoscopic surgery as the assistant surgeon.
* No prior simulation training (mechanical, PC-based or otherwise).

Exclusion Criteria:

* Persons who are not medical students.
* Medical students with prior clinical experience with laparoscopic surgery as the assistant surgeon.
* Medical students with prior simulation training (mechanical, PC-based or otherwise).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-07; Primary Completion 2005-01 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Establish learning curve for each of seven tasks on the simulator. | 6 months
  For each of the module seven modules, the computer automatically measures set parameters. Each measured parameter that is recorded in the simulator will be used in data analysis.

SECONDARY OUTCOMES:
Establish test-retest reliability for each of seven tasks on the simulator. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dennis L Fowler, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States